Study: # 7193 entitled NEUROCOGNITIVE MECHANISMS OF DISULFIRAM TREATMENT OF ALCOHOL USE DISORDER

PI: Nasir Naqvi, MD, PhD

NCT# NCT02735577

Data Analysis Plan created: November 14, 2014

<u>Data Analysis:</u> Functional images will be pre-processed according to standard procedures. A whole-brain general linear model analysis will examine effects of time-point (pre-DIS vs. post-DIS) and cue-type (alcohol vs. food), as well as interaction effects. Psychophysiological interaction analysis will examine cue-elicited functional connectivity between the VS and its inputs from the insula, VMPFC and DLPFC, and how these are changed from pre- to post-DIS. Statistical mediation analyses will determine the extent to which these changes are mediated by the perceived likelihood and salience of the DIS alcohol reaction. Logistic regression analysis will be used to determine whether post-DIS cue-induced VS activity predicts drinking during 1 month of DIS, after controlling for pre-DIS cue-induced VS activity, as well as for AUD severity, motivation, risk-taking, insight and impulsivity.